CLINICAL TRIAL: NCT03117140
Title: A Prospective Triple-masked Randomized Controlled Trial Measuring Analgesia Duration of Dexamethasone, Buprenorphine, or Clonidine With Ropivacaine for Interscalene Nerve Block
Brief Title: Analgesia Duration of Dexamethasone, Buprenorphine, or Clonidine With Ropivacaine for Interscalene Nerve Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melinda Seering (Other)
Responsible Party: Sponsor-Investigator, Melinda Seering, Clinical Assistant Profession, Prinicipal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201304727
Record Dates: First submitted 2017-04-11; First posted 2017-04-17 (Actual); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Anesthesia, Local
Keywords: Brachial Plexus Block; Clonidine; Dexamethasone; Buprenorphine
MeSH Terms: interventions — Ropivacaine; Buprenorphine; Clonidine; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Plain Ropivacaine (Active Comparator): Plain Ropivacaine 0.75%, (225 mg) total volume 32 cc for interscalene block given pre-operatively
  Interventions: Drug: Ropivacaine 0.75%
- Ropivacaine + Buprenorphine (Experimental): A mixture of 0.75% ropivacaine with 300 mcg buprenorphine, total volume 32 cc for interscalene block given pre-operatively
  Interventions: Drug: Ropivacaine 0.75% + 300 mcg Buprenorphine
- Ropivacaine + Clonidine (Experimental): A mixture of 0.75% ropivacaine with 75 mcg clonidine, total volume 32 cc for interscalene block given pre-operatively
  Interventions: Drug: Ropivacaine 0.75% + 75 mcg clonidine
- Ropivaciane + Dexamethasone (Experimental): A mixture of 0.75% ropivacaine with and 8 mg dexamethasone, total volume 32 cc for interscalene block given pre-operatively
  Interventions: Drug: Ropivacaine 0.75% + 8 mg dexamethasone

INTERVENTIONS:
Drug: Ropivacaine 0.75% — Only ropivacaine 0.75% is administered for this arm of the interscalene block
  Other Names: Naropin
  Arms: Plain Ropivacaine
Drug: Ropivacaine 0.75% + 300 mcg Buprenorphine — Ropivacaine 0.75% + 300 mcg Buprenorphine is administered for this arm of the interscalene block
  Other Names: Naropin + Buprenex
  Arms: Ropivacaine + Buprenorphine
Drug: Ropivacaine 0.75% + 75 mcg clonidine — Ropivacaine 0.75% + 75 mcg Clonidine is administered for this arm of the interscalene block
  Other Names: Naropin + Duraclon
  Arms: Ropivacaine + Clonidine
Drug: Ropivacaine 0.75% + 8 mg dexamethasone — Ropivacaine 0.75% + 8 mg Dexamethasone is administered for this arm of the interscalene block
  Other Names: Naropin + Decadron
  Arms: Ropivaciane + Dexamethasone

SUMMARY:
This is a prospective randomized controlled triple-masked study looking at the duration of nerve block analgesia when using the listed adjuvants (dexamethasone, buprenorphine and clonidine) plus ropivacaine versus plain ropivacaine alone.

DETAILED DESCRIPTION:
This is a prospective randomized controlled triple-masked study looking at the duration of nerve block analgesia when using the listed adjuvants (dexamethasone, buprenorphine and clonidine) plus ropivacaine versus plain ropivacaine alone. This will be looked on on patients undergoing painful shoulder surgery in the ambulatory surgery center. Patients will be randomized to one of four groups (1. 0.75% plain ropivacaine. The reference comparator 2. A mixture of 0.75% ropivacaine with 300 mcg buprenorphine 3. A mixture of 0.75% ropivacaine with 75 mcg clonidine 4. A mixture of 0.75% ropivacaine with and 8mg dexamethasone) for their regimen in the interscalene block for their surgery. The patients will then be called within 3 days post-operatively to follow-up. Follow-up data collected will be when did the patient experience return of pain to the operative limb (duration of analgesia), when did the patient experience return of motor function of the operative limb (duration of motor block) and when did the patient experience return of sensation of the operative limb (return of sensory block). All three of these adjuvants have been studied previously and shown to have increased analgesic duration with local anesthesia, but have never had a good comparative study. The mechanism of action of the analgesia for these adjuvants pain relief has never been shown although it is likely a indirect effect as there are animal studies looking at their effect on A and C fibers that did not show those results.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have or are:

  1. Orthopedics service patients having shoulder surgery
  2. ASA(American Society of Anesthesiologists) class I, II, or III.
  3. Patients at least 18 years old but less than 71 years old.
  4. Patients giving informed consent.
  5. Non-Emergency Surgery

     Exclusion Criteria:
* Patients who have or are:

  1. An inability to cooperate during the block placement.
  2. Neuropathy of the planned extremity to block
  3. Diabetes
  4. Documented Kidney Disease
  5. Documented Liver Disease
  6. A lack of or inability to give informed consent.
  7. Currently incarcerated.
  8. Pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-12; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Seering, M.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospital and Clinics, Ambulatory Surgery Clinic, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brummett CM, Williams BA. Additives to local anesthetics for peripheral nerve blockade. Int Anesthesiol Clin. 2011 Fall;49(4):104-16. doi: 10.1097/AIA.0b013e31820e4a49. PMID 21956081
- [Background] Yilmaz-Rastoder E, Gold MS, Hough KA, Gebhart GF, Williams BA. Effect of adjuvant drugs on the action of local anesthetics in isolated rat sciatic nerves. Reg Anesth Pain Med. 2012 Jul-Aug;37(4):403-9. doi: 10.1097/AAP.0b013e3182485965. PMID 22430023
- [Background] Ilfeld BM, Morey TE, Enneking FK. Continuous infraclavicular brachial plexus block for postoperative pain control at home: a randomized, double-blinded, placebo-controlled study. Anesthesiology. 2002 Jun;96(6):1297-304. doi: 10.1097/00000542-200206000-00006. PMID 12170039
- [Background] Ilfeld BM, Morey TE, Thannikary LJ, Wright TW, Enneking FK. Clonidine added to a continuous interscalene ropivacaine perineural infusion to improve postoperative analgesia: a randomized, double-blind, controlled study. Anesth Analg. 2005 Apr;100(4):1172-1178. doi: 10.1097/01.ASN.0000145571.41015.D5. PMID 15781540
- [Background] Ilfeld BM, Morey TE, Wang RD, Enneking FK. Continuous popliteal sciatic nerve block for postoperative pain control at home: a randomized, double-blinded, placebo-controlled study. Anesthesiology. 2002 Oct;97(4):959-65. doi: 10.1097/00000542-200210000-00031. PMID 12357165
- [Background] Ilfeld BM, Vandenborne K, Duncan PW, Sessler DI, Enneking FK, Shuster JJ, Theriaque DW, Chmielewski TL, Spadoni EH, Wright TW. Ambulatory continuous interscalene nerve blocks decrease the time to discharge readiness after total shoulder arthroplasty: a randomized, triple-masked, placebo-controlled study. Anesthesiology. 2006 Nov;105(5):999-1007. doi: 10.1097/00000542-200611000-00022. PMID 17065895
- [Background] White PF, Issioui T, Skrivanek GD, Early JS, Wakefield C. The use of a continuous popliteal sciatic nerve block after surgery involving the foot and ankle: does it improve the quality of recovery? Anesth Analg. 2003 Nov;97(5):1303-1309. doi: 10.1213/01.ANE.0000082242.84015.D4. PMID 14570643
- [Background] Capdevila X, Pirat P, Bringuier S, Gaertner E, Singelyn F, Bernard N, Choquet O, Bouaziz H, Bonnet F; French Study Group on Continuous Peripheral Nerve Blocks. Continuous peripheral nerve blocks in hospital wards after orthopedic surgery: a multicenter prospective analysis of the quality of postoperative analgesia and complications in 1,416 patients. Anesthesiology. 2005 Nov;103(5):1035-45. doi: 10.1097/00000542-200511000-00018. PMID 16249678
- [Background] Saporito A, Sturini E, Petri J, Borgeat A, Aguirre JA. Case report: unusual complication during outpatient continuous regional popliteal analgesia. Can J Anaesth. 2012 Oct;59(10):958-62. doi: 10.1007/s12630-012-9758-9. Epub 2012 Jul 25. PMID 22829027
- [Background] Candido KD, Franco CD, Khan MA, Winnie AP, Raja DS. Buprenorphine added to the local anesthetic for brachial plexus block to provide postoperative analgesia in outpatients. Reg Anesth Pain Med. 2001 Jul-Aug;26(4):352-6. doi: 10.1053/rapm.2001.23931. PMID 11464356
- [Background] Candido KD, Winnie AP, Ghaleb AH, Fattouh MW, Franco CD. Buprenorphine added to the local anesthetic for axillary brachial plexus block prolongs postoperative analgesia. Reg Anesth Pain Med. 2002 Mar-Apr;27(2):162-7. doi: 10.1053/rapm.2002.30671. PMID 11915063
- [Background] Candido KD, Hennes J, Gonzalez S, Mikat-Stevens M, Pinzur M, Vasic V, Knezevic NN. Buprenorphine enhances and prolongs the postoperative analgesic effect of bupivacaine in patients receiving infragluteal sciatic nerve block. Anesthesiology. 2010 Dec;113(6):1419-26. doi: 10.1097/ALN.0b013e3181f90ce8. PMID 21042200
- [Background] Cummings KC 3rd, Napierkowski DE, Parra-Sanchez I, Kurz A, Dalton JE, Brems JJ, Sessler DI. Effect of dexamethasone on the duration of interscalene nerve blocks with ropivacaine or bupivacaine. Br J Anaesth. 2011 Sep;107(3):446-53. doi: 10.1093/bja/aer159. Epub 2011 Jun 14. PMID 21676892
- [Background] Vieira PA, Pulai I, Tsao GC, Manikantan P, Keller B, Connelly NR. Dexamethasone with bupivacaine increases duration of analgesia in ultrasound-guided interscalene brachial plexus blockade. Eur J Anaesthesiol. 2010 Mar;27(3):285-8. doi: 10.1097/EJA.0b013e3283350c38. PMID 20009936
- [Background] Kim YJ, Lee GY, Kim DY, Kim CH, Baik HJ, Heo S. Dexamathasone added to levobupivacaine improves postoperative analgesia in ultrasound guided interscalene brachial plexus blockade for arthroscopic shoulder surgery. Korean J Anesthesiol. 2012 Feb;62(2):130-4. doi: 10.4097/kjae.2012.62.2.130. Epub 2012 Feb 20. PMID 22379567
- [Background] Movafegh A, Razazian M, Hajimaohamadi F, Meysamie A. Dexamethasone added to lidocaine prolongs axillary brachial plexus blockade. Anesth Analg. 2006 Jan;102(1):263-7. doi: 10.1213/01.ane.0000189055.06729.0a. PMID 16368840
- [Background] Casati A, Magistris L, Fanelli G, Beccaria P, Cappelleri G, Aldegheri G, Torri G. Small-dose clonidine prolongs postoperative analgesia after sciatic-femoral nerve block with 0.75% ropivacaine for foot surgery. Anesth Analg. 2000 Aug;91(2):388-92. doi: 10.1097/00000539-200008000-00029. PMID 10910854
- [Background] Couture DJ, Cuniff HM, Maye JP, Pellegrini J. The addition of clonidine to bupivacaine in combined femoral-sciatic nerve block for anterior cruciate ligament reconstruction. AANA J. 2004 Aug;72(4):273-8. PMID 15354916
- [Background] Duma A, Urbanek B, Sitzwohl C, Kreiger A, Zimpfer M, Kapral S. Clonidine as an adjuvant to local anaesthetic axillary brachial plexus block: a randomized, controlled study. Br J Anaesth. 2005 Jan;94(1):112-6. doi: 10.1093/bja/aei009. Epub 2004 Oct 29. PMID 15516351
- [Background] Sripada R, Bowens C Jr. Regional anesthesia procedures for shoulder and upper arm surgery upper extremity update--2005 to present. Int Anesthesiol Clin. 2012 Winter;50(1):26-46. doi: 10.1097/AIA.0b013e31821a0284. PMID 22227421
- [Background] Williams BA. Forecast for perineural analgesia procedures for ambulatory surgery of the knee, foot, and ankle: applying patient-centered paradigm shifts. Int Anesthesiol Clin. 2012 Winter;50(1):126-42. doi: 10.1097/AIA.0b013e31821a00d0. PMID 22227428
- [Background] Williams BA, Hough KA, Tsui BY, Ibinson JW, Gold MS, Gebhart GF. Neurotoxicity of adjuvants used in perineural anesthesia and analgesia in comparison with ropivacaine. Reg Anesth Pain Med. 2011 May-Jun;36(3):225-30. doi: 10.1097/AAP.0b013e3182176f70. PMID 21519308
- [Background] Ahadian FM, McGreevy K, Schulteis G. Lumbar transforaminal epidural dexamethasone: a prospective, randomized, double-blind, dose-response trial. Reg Anesth Pain Med. 2011 Nov-Dec;36(6):572-8. doi: 10.1097/AAP.0b013e318232e843. PMID 22005659
- [Background] Bonhomme V, Doll A, Dewandre PY, Brichant JF, Ghassempour K, Hans P. Epidural administration of low-dose morphine combined with clonidine for postoperative analgesia after lumbar disc surgery. J Neurosurg Anesthesiol. 2002 Jan;14(1):1-6. doi: 10.1097/00008506-200201000-00001. PMID 11773815
- [Background] Vukovic J, Ramakrishnan P, Milan Z. Does epidural clonidine improve postoperative analgesia in major vascular surgery? Med Glas (Zenica). 2012 Feb;9(1):49-55. PMID 22634908
- [Background] Walker SM, Yaksh TL. Neuraxial analgesia in neonates and infants: a review of clinical and preclinical strategies for the development of safety and efficacy data. Anesth Analg. 2012 Sep;115(3):638-62. doi: 10.1213/ANE.0b013e31826253f2. Epub 2012 Jul 13. PMID 22798528
- [Background] Kawamoto S, Tatsumi K, Kataoka T, Kamikawa T, Yanagida T, Mandai R. [Comparison of intrathecal morphine and buprenorphine for postoperative analgesia in cesarean delivery]. Masui. 2011 Aug;60(8):892-6. Japanese. PMID 21861411
- [Background] Modi M, Rastogi S, Kumar A. Buprenorphine with bupivacaine for intraoral nerve blocks to provide postoperative analgesia in outpatients after minor oral surgery. J Oral Maxillofac Surg. 2009 Dec;67(12):2571-6. doi: 10.1016/j.joms.2009.07.014. PMID 19925973
- [Background] Ip VH, Tsui BC. Practical concepts in the monitoring of injection pressures during peripheral nerve blocks. Int Anesthesiol Clin. 2011 Fall;49(4):67-80. doi: 10.1097/AIA.0b013e31821775bc. No abstract available. PMID 21956078
- [Background] Tsui BC, Li LX, Pillay JJ. Compressed air injection technique to standardize block injection pressures. Can J Anaesth. 2006 Nov;53(11):1098-102. doi: 10.1007/BF03022877. PMID 17079636
- [Background] Auroy Y, Benhamou D, Bargues L, Ecoffey C, Falissard B, Mercier FJ, Bouaziz H, Samii K. Major complications of regional anesthesia in France: The SOS Regional Anesthesia Hotline Service. Anesthesiology. 2002 Nov;97(5):1274-80. doi: 10.1097/00000542-200211000-00034. PMID 12411815
- [Background] Neal JM, Bernards CM, Hadzic A, Hebl JR, Hogan QH, Horlocker TT, Lee LA, Rathmell JP, Sorenson EJ, Suresh S, Wedel DJ. ASRA Practice Advisory on Neurologic Complications in Regional Anesthesia and Pain Medicine. Reg Anesth Pain Med. 2008 Sep-Oct;33(5):404-15. doi: 10.1016/j.rapm.2008.07.527. PMID 18774509
- [Background] Laur JJ, Chehade JM, Merrill DG. Managing neural dysfunction after regional anesthesia: experience in a walk-in follow-up clinic. Int Anesthesiol Clin. 2011 Summer;49(3):44-55. doi: 10.1097/AIA.0b013e318217fe85. No abstract available. PMID 21697669

RESULTS

PARTICIPANT FLOW:
Groups:
- Plain Ropiviciane: Plain Ropivicaine 0.75%, (225 mg) total volume 32 cc for interscalene block given pre-operatively
  Ropivicaine 0.75%: Only ropivicaine 0.75% is administered for this arm of the interscalene block
- Ropiviciane + Buprenorphine: A mixture of 0.75% ropivacaine with 300 mcg buprenorphine, total volume 32 cc for interscalene block given pre-operatively
  Ropivicaine 0.75% + 300 mcg Buprenorphine: Ropivicaine 0.75% + 300 mcg Buprenorphine is administered for this arm of the interscalene block
- Ropivicaine + Clonidine: A mixture of 0.75% ropivacaine with 75 mcg clonidine, total volume 32 cc for interscalene block given pre-operatively
  Ropivicaine 0.75% + 75 mcg clonidine: Ropivicaine 0.75% + 75 mcg Clonidine is administered for this arm of the interscalene block
- Ropiviciane + Dexamethasone: A mixture of 0.75% ropivacaine with and 8 mg dexamethasone, total volume 32 cc for interscalene block given pre-operatively
  Ropivicaine 0.75% + 8 mg dexamethasone: Ropivicaine 0.75% + 8 mg Dexamethasone is administered for this arm of the interscalene block
Period: Overall Study
Arm/Group | Plain Ropiviciane | Ropiviciane + Buprenorphine | Ropivicaine + Clonidine | Ropiviciane + Dexamethasone
Started | 40 | 40 | 40 | 40
Completed | 40 | 40 | 40 | 40
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ropivacaine + Dexamethasone: A mixture of 0.75% ropivacaine with and 8 mg dexamethasone, total volume 32 cc for interscalene block given pre-operatively
  Ropivacaine 0.75% + 8 mg dexamethasone: Ropivacaine 0.75% + 8 mg dexamethasone is administered for this arm of the interscalene block
- Total: Total of all reporting groups
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone | Total
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 38 | 39 | 40 | 154
  >=65 years | 3 | 2 | 1 | 0 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.38 (14.39) | 44.8 (14.2) | 43.1 (14.74) | 42.3 (13.71) | 43.89 (14.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 7 | 9 | 40
  Male | 25 | 31 | 33 | 31 | 120
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ASA (American Society of Anesthesiolgy) Classification system [Count of Participants; unit: Participants] — I-a normal healthy patient II- a patient with mild systemic disease III-a patient with severe systemic disease
  Participants
    ASA classification I | 13 | 14 | 15 | 17 | 59
    ASA classification II | 23 | 24 | 18 | 21 | 86
    ASA classification III | 4 | 2 | 7 | 2 | 15
Weight [Mean (Standard Deviation); unit: kilograms] | 98.82 (22.71) | 98.13 (21.47) | 99.78 (25.95) | 95.63 (21.41) | 98.09 (22.79)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Analgesia
Description: Patients are called 1-3 days post-operatively to assess when the analgesia of their nerve block wore off
Time Frame: 1-3 days post-operative
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
Number analyzed (Participants) | 40 | 40 | 40 | 40
minutes | 911 [652 to 1300] | 1026.5 [756.5 to 1392.5] | 1181 [880.5 to 1528.5] | 982 [799 to 1270]

2. Secondary Outcome: Block Set up Time
Description: Patients are assessed from needle removal to when they are no longer able to feel cold on the blocked extremity
Time Frame: Day one
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
Number analyzed (Participants) | 40 | 40 | 40 | 40
minutes | 6 [3 to 9] | 3 [3 to 6] | 6 [3 to 6] | 4.5 [3 to 10.5]

3. Secondary Outcome: Sensory Duration of Block
Description: Patients are called 1-3 days post-operatively to assess when the sensory component of their nerve block wore off
Time Frame: Day 1-3
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
Number analyzed (Participants) | 40 | 40 | 40 | 40
minutes | 923.5 [652 to 1304] | 982 [705 to 1189] | 940.5 [736.5 to 1234] | 1066 [797 to 1240]

4. Secondary Outcome: Patient Reporting Vomiting at Home
Description: Patients are called 1-3 days post-operatively to assess if they had any side effects of the adjuvants such as nausea, vomiting or itching. There blood pressure is looked at pre-op and compared to post-op. Any prolonged PACU (Post Anesthesia Care Unit) stay for sedation is recorded.
Time Frame: 1-3 days
Population: 1 patient in the Plain Ropivacaine group and the Ropivacaine and Buprenorphine group did not complete the survey about vomiting at home and therefore was not included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
Number analyzed (Participants) | 39 | 39 | 40 | 40
Participants | 0 | 3 | 2 | 1

5. Secondary Outcome: Number of Patients Vomiting in the PACU (Post-Anesthesia Care Unit)
Description: Vomiting in PACU (Post-Anesthesia Care Unit) for patients was looked at
Time Frame: Post-op Day 0 (Baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
Number analyzed (Participants) | 40 | 40 | 40 | 40
Participants | 0 | 1 | 0 | 0

6. Secondary Outcome: Number of Patients Reporting Nausea at Home
Description: as for outcome 4
Time Frame: 1-3 days
Population: 1 patient in the Plain Ropivacaine group and the Ropivacaine and Buprenorphine group did not complete the survey about nausea at home and therefore was not included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
Number analyzed (Participants) | 39 | 39 | 40 | 40
Participants | 4 | 9 | 2 | 3

7. Secondary Outcome: Number of Patients Reporting Nausea in the PACU
Description: PACU (Post-Anesthesia Care Unit) assessment of nausea
Time Frame: Post-op day 0 (Baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
Number analyzed (Participants) | 40 | 40 | 40 | 40
Participants | 4 | 9 | 2 | 9

8. Secondary Outcome: Motor Duration of Block
Description: Patients are called 1-3 days post-operatively to assess when motor component of their nerve block wore off
Time Frame: Day 1-3
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Plain Ropivacaine: Plain Ropivacaine 0.75%, (225 mg) total volume 32 cc for interscalene block given pre-operatively
  Ropivacaine 0.75%: Only ropivicaine 0.75% is administered for this arm of the interscalene block
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
Number analyzed (Participants) | 40 | 40 | 40 | 40
minutes | 1120 [748 to 1484] | 1198 [835 to 1406] | 1090 [829 to 1526] | 1143.5 [949.5 to 1356.5]

9. Secondary Outcome: Number of Patients With Blood Pressure (BP) Changes in the PACU
Description: Blood pressure changes in PACU (Post-Anesthesia Care Unit) for patients was looked at
Time Frame: Post-op Day 0 (baseline)
Population: 1 patient in Ropivacaine and Buprenorphine group did get data for the BP changes in the PACU for the study so therefore was not included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
Number analyzed (Participants) | 40 | 39 | 40 | 40
Participants | 8 | 3 | 7 | 2

10. Secondary Outcome: Number of Patient With Blood Pressure Changes in the Second Stage Recovery Area
Description: Blood pressure changes in Second Stage Recovery Area for patients was looked at
Time Frame: Post-op Day 0 (baseline)
Population: 1 patient in Ropivacaine and Buprenorphine group did not have blood pressure data obtained in the second stage area so therefore was not included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
Number analyzed (Participants) | 40 | 39 | 40 | 40
Participants | 5 | 1 | 5 | 0

11. Secondary Outcome: Pain Score Reported by Patients at First Phone Call
Description: Patients are called 1-3 days post-operatively to assess pain. Pain score is 0-10 scale with 0 is no pain and 10 is most severe pain.
Time Frame: Day 1-3
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
Number analyzed (Participants) | 40 | 40 | 40 | 40
units on a scale | 4 [3 to 5] | 3 [2 to 5] | 4 [2 to 5.5] | 3 [2 to 4.5]

12. Secondary Outcome: Number of Patients Reporting Itching in the PACU
Description: Patients itching was assessed post-op in the PACU.
Time Frame: Post-op day 0 (baseline)
Population: 1 patient in the Ropivacaine and Buprenorphine group did not obtain data on the itching in the PACU therefore was not included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
Number analyzed (Participants) | 40 | 39 | 40 | 40
Participants | 5 | 2 | 6 | 3

13. Secondary Outcome: Number of Patients Reporting Itching at Home
Description: as for outcome 4
Time Frame: 1-3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
Number analyzed (Participants) | 40 | 40 | 40 | 40
Participants | 1 | 2 | 2 | 0

14. Other Pre Specified Outcome: Surgical Position
Description: Surgical position was recorded
Time Frame: Post-op Day 0 (Baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
Number analyzed (Participants) | 40 | 40 | 40 | 40
Participants
  Beach Chair | 38 | 31 | 31 | 32
  Lateral | 2 | 6 | 7 | 6
  Supine | 0 | 3 | 2 | 2

15. Other Pre Specified Outcome: Surgical Length
Description: Surgical length was recorded
Time Frame: Post op Day 0 (Baseline)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
Number analyzed (Participants) | 40 | 40 | 40 | 40
minutes | 68.5 [45 to 94] | 65 [49 to 87.5] | 73.5 [56 to 101] | 71 [47.5 to 117]

ADVERSE EVENTS:
Time Frame: The adverse advents data was collected from Day 1 until Day 3 when the phone call was made. We do have a post-block clinic where patients with adverse events post-block are seen. None from the study were seen here.
Arm/Group | Plain Ropivacaine | Ropivacaine + Buprenorphine | Ropivacaine + Clonidine | Ropivacaine + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-06-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT03117140/Prot_SAP_000.pdf